CLINICAL TRIAL: NCT07259044
Title: Global Strategies, Local Impact: Testing Scalable Caregiver Interventions for Autism in Low-Resource Health Systems
Brief Title: Testing Scalable Caregiver Interventions for Autism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Moi University (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Megan Song McHenry, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 96463446
Record Dates: First submitted 2025-09-24; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder; Autism; ASD
Keywords: Caregiver Intervention; Training; Children; Low Resource; Disability; Early Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: At each site, groups will be randomly assigned to be led by either trained professionals (e.g., occupational therapists or special education teachers) or peer facilitators (caregivers of children with autism trained in the curriculum).
Who Masked: Outcomes Assessor
Masking Description: Data collectors will be masked to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Professional-led Caregiver Groups (Experimental)
  Interventions: Behavioral: Professionally-facilitated groups
- Peer-facilitated Caregiver Groups (Experimental)
  Interventions: Behavioral: Peer-facilitated groups
- Waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: Professionally-facilitated groups — A group-based caregiver ASD intervention will be delivered through two distinct implementation strategies led by trained therapists or teachers using a structured 10-week in-person curriculum at the MTRH campus and virtually in the US.
  Arms: Professional-led Caregiver Groups
Behavioral: Peer-facilitated groups — A group-based caregiver ASD intervention will be delivered through two distinct implementation strategies led by trained caregivers of children with ASD who deliver the same core curriculum with flexibility in timing and location, provided that all content is completed within four months.
  Arms: Peer-facilitated Caregiver Groups

SUMMARY:
Autism spectrum disorder affects 1-2% of children worldwide, yet access to quality care remains limited, especially in underserved communities. Families face systemic barriers such as workforce shortages, high caregiver stress, and a lack of culturally appropriate services.

To address these gaps, researchers developed a group-based caregiver training program to improve caregiver well-being and child communication and behavior. Successfully piloted in rural U.S. communities and western Kenya through the AMPATH Program, the intervention showed promising results in reducing caregiver stress and autism severity.

Building on this success, a new study will evaluate two delivery models-professionally-led and peer-led-using a rigorous effectiveness-implementation trial. The project applies a reciprocal innovation approach, using insights from Kenya to inform U.S. strategies for scaling community-based autism support.

The long-term goal is to reduce disparities in autism care by creating scalable, low-cost, caregiver-driven models. A Community Advisory Panel will guide the research to ensure relevance and impact. This initiative represents a transformative step toward equitable autism services across global and U.S. settings.

DETAILED DESCRIPTION:
Autism spectrum disorder is a common neurodevelopmental disability affecting 1-2% of children worldwide. While early intervention is critical for improving outcomes, access to quality services remains severely limited. Families in low-resource settings, both globally and within the U.S, face systemic barriers including workforce shortages, high caregiver burden, and limited culturally appropriate services. There is a critical need for scalable low-cost interventions to support children with autism and their families in communities where robust systems of care are absent.

To address this gap, researchers developed a group-based caregiver training intervention to support caregiver well-being and communication and behavior in children with autism. Piloted successfully in rural U.S. and western Kenya through the Academic Model Providing Access to Healthcare (AMPATH) Program, the intervention demonstrated feasibility, acceptability, and improvements in caregiver stress, child communication and behavior scores, and autism severity scores. Building on this foundation, researchers propose a Hybrid Type 2 effectiveness-implementation trial to rigorously evaluate both the intervention's effectiveness of improving child and caregiver outcomes and the implementation strategies needed for sustainable scale-up across health systems. The researchers embed a reciprocal innovation approach, leveraging insights from Kenya to inform U.S. communities facing similar challenges. Specifically, lessons learned from scaling peer-led delivery models in Kenya, where scare autism resources exist, will directly inform efforts to expand community-based autism support services in underserved areas of the U.S., where similar implementation challenges persist and services are variable.

The long-term goal is to reduce disparities in autism care and outcomes by developing scalable, community-driven caregiver support models. The researchers will bring together a Community Advisory Panel to ensure clinical and scientific rigor to maximize translation of findings. The overall objective of this study is to evaluate the effectiveness and implementation outcomes, including cost-effectiveness, of professional-led versus peer-led caregiver support for children with autism in Kenya, and to leverage lessons learned to reciprocally pilot-test the peer-led intervention in the U.S. To achieve this objective, the investigators propose the following Aims:

Aim 1: Evaluate the effectiveness of a group-based caregiver training program on caregiver and child outcomes in Kenya. Approach: Investigators will conduct a cluster randomized trial comparing two delivery strategies for a caregiver-focused autism intervention, either (1) structured delivery by trained professionals (e.g. therapists, teachers) using standardized scripts and materials, or (2) peer-led delivery by trained caregivers of children with autism with guided instruction; with a staggered wait-list control. Outcomes will be assessed for caregivers (quality of life (QOL), stress/burden, depressive symptoms) and children (functional communication, behavioral challenges, QOL) at enrollment, pre-/post-intervention, and 3-month follow-up. The investigators hypothesize that the caregiver training program will lead to sustained improvements in caregiver and child outcomes overall, and peer-led delivery of the intervention will be non-inferior to professional-led delivery, supporting its potential for scalability and sustainability.

Aim 2: Determine and compare key implementation outcomes, including cost-effectiveness, between two intervention delivery strategies-in-person, professional- vs. peer-led caregiver groups. Approach: Guided by the Consolidated Framework for Implementation Research (CFIR), investigators will use mixed-methods to analyze implementation outcomes of both intervention delivery strategies, including cost-effectiveness, fidelity, acceptability, feasibility, among others. A community advisor board will guide interpretation. The investigators hypothesize that while acceptability and appropriateness may be similar between the two delivery strategies, the trained peer-led delivery will demonstrate greater feasibility and lower cost, providing key insights to support piloting and scale-up in the U.S.

Aim 3: Optimize and pilot a peer-led autism caregiver intervention in the U.S., measuring key effectiveness and implementation outcomes to support scale-up in U.S. underserved settings. Approach: The investigators will use an implementation science and ecological validity framework adaptation process to revise the peer-led program for delivery in the U.S. Building on lessons from the Kenya, trained peers will deliver the adapted pilot program in Virginia. The investigators will use an explanatory sequential mixed-methods approach to evaluate effectiveness and implementation outcomes. The investigators hypothesize that the peer-led model will be feasible, acceptable, and delivered with high fidelity in U.S. under-served settings, with effectiveness, demonstrating reciprocal innovation from Kenya to the U.S. and provide key foundational insights for future scale-up.

This study's innovation lies in that it will be among the first rigorous evaluations of a scalable, caregiver-mediated autism intervention in low-resourced settings using an implementation science framework. Lessons learned from scaling peer-led delivery models in Kenya, where children receive very few services for autism, can directly inform efforts to expand community-based autism support services in underserved areas of the U.S., where similar implementation challenges persist and services are variable, for significant impact. This bidirectional learning model represents a transformative approach to developing and delivering scalable, equitable autism care throughout the U.S. and globally.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver is willing to participate
* Caregiver speaks either Swahili or English
* Child is between 2 and 8 years of age
* Child presents with concerns suggestive of autism

Exclusion Criteria:

* The caregiver declines to participate
* The child has significant vision or hearing impairment
* The child is not primarily cared for by the enrolled caregiver

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Family Burden and Stress | Baseline and 3 months
  Change in caregiver-reported burden and stress levels from baseline to 3 months, measured using the Caregiver Self-Assessment Questionnaire developed by the American Medical Association. This 18-item tool includes 16 yes/no items assessing emotional and physical strain, one item rating stress on a scale from 1 (no stress) to 10 (high stress), and one item comparing current health to health one year ago. Higher scores indicate greater caregiver burden and stress.
Autism Impact Measure (AIM) | Baseline and 3 months
  Change in caregiver-reported communication and symbolic behavior from baseline to 3 months, measured using the Autism Impact Measure (AIM), which integrates domains from the Communication and Symbolic Behavior Scale (CSBS). The AIM is a validated caregiver-report tool assessing autism-related behaviors across five domains, including communication and social reciprocity. The CSBS is a norm-referenced, standardized instrument that evaluates early communication development through 22 rating scales grouped into seven clusters: communicative functions, gestural and vocal means, verbal means, reciprocity, social-affective signaling, and symbolic behavior. Higher AIM scores indicate greater autism-related impact.

SECONDARY OUTCOMES:
Quality of Life in Caregivers | Baseline and 3 months
  Change in caregiver-reported quality of life from baseline to 3 months, measured using the Quality of Life - Family Version instrument developed by Betty Ferrell, PhD. This 37-item ordinal scale assesses quality of life across four domains for family members caring for a patient. Each item is rated from 0 (worst outcome) to 10 (best outcome), with several items reverse-scored. Subscale scores are calculated by averaging items within each domain. Higher overall scores indicate better caregiver quality of life.
Quality of Life in Children | Baseline and 3 months
  Change in caregiver-reported quality of life for children from baseline to 3 months, measured using the Pediatric Quality of Life Inventory (PedsQL) Generic Core Scales. This 23-item instrument assesses physical, emotional, social, and school functioning across four multidimensional scales and three summary scores. It is developmentally appropriate for ages 2-18 and includes both child self-report (ages 5-18) and parent proxy-report (ages 2-18). Scores range from 0 to 100, with higher scores indicating better quality of life.
Parenting Stress Index | Baseline and 3 months
  Change in parenting stress from baseline to 3 months, measured using the Parenting Stress Index-Short Form (PSI-SF). The PSI-SF total score ranges from 36 to 180, with higher scores indicating greater parenting stress and a worse outcome. Each of the 36 items is rated on a 5-point Likert scale, and the measure includes three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child.
Depressive Symptoms in Caregivers | Baseline and 3 months
  Change in caregiver depressive symptoms from baseline to 3 months, measured using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 score ranges from 0 to 27, with higher scores indicating more severe depression and a worse outcome. Each item is scored from 0 (not at all) to 3 (nearly every day).
Child Behavior Checklist (CBCL) | Baseline and 3 months
  Change in child behavior scores from baseline to 3 months, as reported by caregivers using the Child Behavior Checklist (CBCL). The CBCL is part of the Achenbach System of Empirically Based Assessment and evaluates behavioral and emotional problems in children. Caregivers rate behaviors on a 3-point scale: 0 ("Not True"), 1 ("Somewhat or Sometimes True"), and 2 ("Very True or Often True"). Raw scores are converted to T-scores ranging from 0 to 100. Higher T-scores indicate greater behavioral or emotional problems and a worse outcome.
Delivery Method Comparison: Peer-led vs Professional-led Intervention | 3 months
  Comparison of effectiveness between peer-led and professional-led delivery of the caregiver autism intervention using a non-inferiority approach. The estimand is the mean difference in baseline-adjusted communication scores at 3 months, measured using the Communication and Symbolic Behavior Scale (CSBS). The CSBS is a norm-referenced, standardized instrument that evaluates early communication development across 22 rating scales grouped into seven clusters: communicative functions, gestural and vocal means, verbal means, reciprocity, social-affective signaling, and symbolic behavior. Higher scores indicate more advanced communication skills and a better outcome.
Incremental Cost-Effectiveness Ratio (ICER) | 3 months
  Effectiveness and cost will be analyzed jointly using multilevel models with random effects for site and group, and incremental cost-effectiveness ratios (ICERs) will be computed. Net Monetary Benefit (NMB) mixed-effect regressions will allow formal testing of heterogeneity (e.g., baseline severity of autism, living condition, caregiver education and other socioeconomic factors). Uncertainty will be assessed using clustered bootstraps and cost-effectiveness acceptability curves (CEACs).

OTHER OUTCOMES:
Acceptability of Intervention | Post-intervention (6 months)
  Assessed using the Acceptability of Intervention Measure (AIM) and items aligned with the Theoretical Framework of Acceptability (TFA). The AIM is a 4-item scale rated from 1 ("completely disagree") to 5 ("completely agree"), total score range 4-20; higher scores indicate greater acceptability. Supplementary qualitative interviews will be coded using a deductive framework based on CFIR and Proctor's IOF to explore perceived acceptability and inform program adaptation.
Feasibility of Intervention - Quantitative Assessment | Post-intervention (6 months)
  Feasibility of the caregiver autism intervention, assessed using the Feasibility of Intervention Measure (FIM). The FIM is a validated 4-item scale designed to assess the extent to which an intervention can be successfully used or carried out within a given setting. Each item is rated on a 5-point Likert scale from 1 ("completely disagree") to 5 ("completely agree"), yielding a total score range of 4 to 20. Higher scores indicate greater perceived feasibility and a better outcome.
Feasibility of Intervention - Qualitative Assessment | Post-intervention (6 months)
  Feasibility of the caregiver autism intervention, assessed through semi-structured qualitative interviews with caregivers and facilitators. Transcripts will be coded using a deductive codebook aligned with the Consolidated Framework for Implementation Research (CFIR) and constructs from Proctor's Implementation Outcomes Framework (IOF). Thematic analysis will identify perceived acceptability, appropriateness, feasibility, reach, barriers, facilitators, and recommended refinements. Findings will be summarized using a joint diagram supported by illustrative quotes.
Fidelity of Intervention Delivery | 10 weeks
  Fidelity of intervention delivery assessed through audio-recorded sessions scored using a standardized fidelity rubric. The rubric evaluates facilitator adherence to core curriculum components, delivery quality, and responsiveness. Fidelity metrics are informed by prior implementation of the Pepea Pamoja and Takia programs. Scores will be aggregated across sessions to produce a mean fidelity score per facilitator. Curriculum adaptations will be documented, and facilitator training will include competency checklists, booster trainings, and structured feedback meetings to support fidelity.
Reach of Intervention | Enrollment through 6-month follow-up
  Assessed using eligibility and retention data, including proportion of eligible caregivers who enrolled and completed the intervention.
Appropriateness of Intervention - Quantitative Assessment Using the Implementation Appropriateness Measure | Post-intervention (6 months)
  Appropriateness of the caregiver autism intervention, assessed using the Implementation Appropriateness Measure (IAM). The IAM is a validated 4-item scale designed to assess the perceived fit, relevance, or compatibility of an intervention for a specific setting or population. Each item is rated on a 5-point Likert scale from 1 ("completely disagree") to 5 ("completely agree"), yielding a total score range of 4 to 20. Higher scores indicate greater perceived appropriateness and a better outcome.
Appropriateness of Intervention - Qualitative Assessment | Post-intervention (6 months)
  Appropriateness of the caregiver autism intervention, assessed through semi-structured qualitative interviews with caregivers and facilitators. Transcripts will be analyzed thematically using a deductive codebook informed by implementation science frameworks, including constructs from the Implementation Outcomes Framework (IOF). Themes will include perceived fit, relevance, and contextual compatibility, supported by illustrative quotes.
Reasons for Attrition | At time of participant withdrawal (if applicable), up to 6 months post-enrollment
  Exit interviews conducted with caregivers who discontinue participation to identify barriers to retention.

CONTACTS AND LOCATIONS:
Overall Officials: Eren Oyungu, MBChB, Principal Investigator — Moi University; Megan S. McHenry, MD, MS, Principal Investigator — Indiana University
Locations (2):
- University of Virginia (Virtual), Charlottesville, Virginia, United States
- Moi Teaching and Referral Hospital, Eldoret, Kenya

REFERENCES:
- [Background] Varni JW. PedsQL™ (Pediatric Quality of Life Inventory™). James W. Varni, Ph.D. Accessed September 18, 2025, https://www.pedsql.org
- [Background] Ferrell BRaG, Marcia. Quality of Life - Family Version. City of Hope National Medical Center and Beckman Research Institute. Accessed September 18, 2025, https://www.cityofhope.org/sites/www/files/2022-06/1431763601545-qol-family%20%282%29.pdf
- [Background] American Psychological Association. Caregiver Self-Assessment Questionnaire. American Psychological Association. Accessed September 18, 2025, https://www.apa.org/pi/about/publications/caregivers/practice-settings/assessment/tools/self-assessment
- [Background] Mwangi P, Nyongesa MK, Koot HM, Cuijpers P, Newton CRJC, Abubakar A. Validation of a Swahili version of the 9-item Patient Health Questionnaire (PHQ-9) among adults living with HIV compared to a community sample from Kilifi, Kenya. J Affect Disord Rep. 2020 Dec;1:100013. doi: 10.1016/j.jadr.2020.100013. PMID 33313580
- [Background] Wetherby AMaP, Barry M. CSBS™ - Communication and Symbolic Behavior Scales. Brookes Publishing Co. Accessed September 18, 2025, https://brookespublishing.com/product/csbs
- [Background] Rutter MB, Anthony; & Lord, Catherine. Social Communication Questionnaire (SCQ®). Western Psychological Services (WPS). Accessed September 18, 2025, https://www.wpspublish.com/scq-social-communication-questionnaire.html
- [Background] Achenbach TM. Child Behavior Checklist for Ages 6-18 (CBCL/6-18). ASEBA, University of Vermont. Accessed September 18, 2025, https://aseba.org/wp-content/uploads/2019/02/schoolagecbcl.pdf
- [Background] Mazurek MO, Carlson C, Baker-Ericzen M, Butter E, Norris M, Barr C, Kanne S. The Autism Impact Measure (AIM): Examination of Sensitivity to Change. Autism Res. 2020 Nov;13(11):1867-1879. doi: 10.1002/aur.2397. Epub 2020 Oct 1. PMID 33001561